CLINICAL TRIAL: NCT05243511
Title: "PROSPER-FM": Prospective Study to Evaluate a Digital Regimen for Fibromyalgia Management
Brief Title: Prospective Study to Evaluate a Digital Regimen for Fibromyalgia Management
Acronym: PROSPER-FM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Swing Therapeutics, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Swing-005
Record Dates: First submitted 2022-02-07; First posted 2022-02-17 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-02

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Digital Acceptance and Commitment Therapy (ACT) Arm (Active Comparator)
  Interventions: Device: Digital ACT
- Digital Symptom Tracker (Active Comparator)
  Interventions: Other: Digital Symptom Tracker

INTERVENTIONS:
Device: Digital ACT — Participants in this arm receive Digital ACT as well as standard of care.
  Arms: Digital Acceptance and Commitment Therapy (ACT) Arm
Other: Digital Symptom Tracker — Participants in this arm complete a digital symptom and function tracker and monitor, are provided access to digital fibromyalgia and health education, and receive standard of care.
  Arms: Digital Symptom Tracker

SUMMARY:
PROSPER-FM is a multi-center, randomized, non-significant risk device study to evaluate the safety and efficacy of two digital therapy smartphone applications in participants with fibromyalgia. Eligible participants are randomized (1:1) to either the Digital Acceptance and Commitment Therapy (Digital ACT) group or the Digital Symptom Tracker group and receive assigned therapy for 12 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

1. Participant is 22 to 75 years of age, inclusive
2. Participant has a diagnosis of primary FM as defined by the 2016 American College of Rheumatology Preliminary Diagnostic Criteria for FM
3. Participants with ongoing treatments should be on stable therapy for 30 days prior to screening appointment.
4. Participant is capable of reading and understanding English and has provided written informed consent to participate.

Key Exclusion Criteria:

1. Lifetime history of bipolar or other psychotic disorder
2. Severe depression at screening (measured by BDI-II)
3. The participant is at increased risk of suicide on the basis of the investigator's judgment or the Columbia-Suicide Severity Rating Scale ("C-SSRS")
4. Participant has any other disease or medical condition that, in the opinion of the Investigator or Sponsor, could endanger the participant, interfere with the evaluation of the study device's efficacy or safety, or compromise the participant's ability to comply with/complete the study.

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2022-02-08 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Patient Global Impression of Change (PGIC) response rate | Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Michael Gendreau, MD, Study Chair — Consulting Chief Medical Officer; Lesley Arnold, MD, Principal Investigator — Study Principal Investigator
Locations (25):
- United States (25):
  - Site #37, Covina, California
  - Site #15, Oceanside, California
  - Site #31, San Bernardino, California
  - Site #38, Thousand Oaks, California
  - Site #36, Tujunga, California
  - Site #35, Whittier, California
  - Site #13, Orlando, Florida
  - Site #33, St. Petersburg, Florida
  - Site #25, Atlanta, Georgia
  - Site #21, Covington, Louisiana
  - Site #20, New Orleans, Louisiana
  - Site #22, Prairieville, Louisiana
  - Site #39, Chestnut Hill, Massachusetts
  - Site #24, Ocean Springs, Mississippi
  - Site #34, Brooklyn, New York
  - Site #32, Scarsdale, New York
  - Site #12, Williamsville, New York
  - Site #27, Fargo, North Dakota
  - Site #14, Cincinnati, Ohio
  - Site #28, Dayton, Ohio
  - Site #23, Tulsa, Oklahoma
  - Site #16, Allentown, Pennsylvania
  - Site #29, Austin, Texas
  - Site #26, McKinney, Texas
  - Site #30, Pflugerville, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gendreau RM, McCracken LM, Williams DA, Luciano JV, Dai Y, Vega N, Ghalib Z, Guthrie K, Kraus AC, Rosenbluth MJ, Vaughn B, Zomnir JM, Reddy D, Chadwick AL, Clauw DJ, Arnold LM. Self-guided digital behavioural therapy versus active control for fibromyalgia (PROSPER-FM): a phase 3, multicentre, randomised controlled trial. Lancet. 2024 Jul 27;404(10450):364-374. doi: 10.1016/S0140-6736(24)00909-7. Epub 2024 Jul 8. PMID 38991582